CLINICAL TRIAL: NCT03490656
Title: Assessment of Investigational Magnetic Resonance Imaging and Post-Processing Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RP0688/2013H0304
Record Dates: First submitted 2018-02-22; First posted 2018-04-06 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: MRI Imaging
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Healthy volunteer population (Experimental)
  Interventions: Diagnostic Test: MRI Scan - not in addition to standard of care
- Patient population (Experimental)
  Interventions: Diagnostic Test: MRI Scan - in addition to standard of care

INTERVENTIONS:
Diagnostic Test: MRI Scan - in addition to standard of care — Up to 3 Tesla (T) MRI
  Arms: Patient population
Diagnostic Test: MRI Scan - not in addition to standard of care — Up to 3 Tesla (T) MRI
  Arms: Healthy volunteer population

SUMMARY:
The goals of this study are to (1) develop and optimize MRI acquisition and post-processing techniques and (2) to generate preliminary and comparative data on sequences for potential clinical trials.

DETAILED DESCRIPTION:
This prospective study will utilize investigational MRI sequences both in a volunteer population as well as in patients in addition to standard of care MR imaging to develop and optimize MRI sequence post-processing techniques as well as to generate preliminary and comparative data for potential clinical trials. These post-processing techniques include but are not limited to visual inspection of image quality and known anatomy, semi-quantitative analysis including the use of rating schemes, signal-to-noise-ratios and contrast-to-noise-ratios measurements for quantitative assessment, standard fitting procedures for measuring MRI parameters, and using various published methods for image post-processing. The MRI methodologies we plan to use as part of this study will allow us to obtain morphological, functional and molecular information. For the patient population: Patients receiving a standard of care 1.5 or 3T MRI will be asked by study personnel if they are interested in undergoing additional investigational imaging sequences after their standard of care imaging. If the patient agrees, he/she will remain in the same position on the MRI scanner for up to an additional 30 minutes while more images are obtained. Each patient will be imaged for no longer than 2 hours (standard of care imaging and additional investigational imaging). A routine clinical report will be generated for the clinically indicated MRI by a radiologist. Once this routine clinical MRI scan is dictated and finalized, a study team member will obtain the report via IHIS and manually remove all identifiers. This report is being obtained for comparative purposes. All the data being compared will be coded using a unique study number. For the volunteer population: Healthy volunteers recruited through the OSU Wexner Medical Center or accompanying patients to their standard of care imaging appointments at The Wright Center of Innovation will be asked by study personnel if they are interested in undergoing investigational MR imaging sequences. If the volunteer agrees, he/she will be imaged on the MRI scanner for up to 60 minutes while images are obtained. Other than the participant signing the informed consent form, no participant information or protected health information (PHI) will be recorded. Following the informed consent authorization, the participant's name will be coded using a unique study number.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers greater than or equal to 18 years of age
* Patients receiving a standard of care 1.5 or 3T MRI at The Ohio State University
* Healthy volunteers that feel comfortable receiving an investigational mRI

Exclusion Criteria:

* Participants with a contraindication to MRI. Such contraindications include, but are not limited to: pacemaker, metallic cardiac valve(s), magnetic material such as surgical clips, tattoos, implanted electronic infusion pumps or any other condition that would interfere with the MRI, a stent somewhere, a history of allergic reaction to any metals
* Participants that experience claustrophobia, anxiety and/or vertigo when moved inside the scanner
* Participants with vital signs outside of normal range
* Prisoners
* Subjects incapable of giving informed written consent
* Participants who are pregnant, healthy volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Image quality | through study completion, an average of 1-3 years
  assessed by blinded readers
Artifacts | through study completion, an average of 1-3 years
  assessed by blinded readers
Lesion detectability | through study completion, an average of 1-3 years
  assessed by blinded readers
Image noise | through study completion, an average of 1-3 years
  assessed region of interest over target tissue and background

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Knopp, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT03490656/Prot_000.pdf